CLINICAL TRIAL: NCT06069700
Title: Effectiveness of Targeted Individualized Multi-modal Treatments in Adults Suffering From Persistent Concussion Symptoms as Compared to Usual Care
Brief Title: Effectiveness of Rehabilitation in Adults Suffering From Persistent Concussion Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: NeuroCatch Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 22-5560
Record Dates: First submitted 2023-09-22; First posted 2023-10-06 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-03

CONDITIONS: Postconcussion Syndrome; Mild Traumatic Brain Injury
MeSH Terms: conditions — Post-Concussion Syndrome; Brain Concussion

STUDY DESIGN:
Intervention Model Description: Randomized cas-crossover clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Individualized care program (Experimental): Participants in the individualized care stream, will be provided reassurance and psychoeducation via the bio-psycho-social model on understanding persistent symptoms consistent with usual care. Additionally, they will be afforded up to 12 treatments over the course of 6-weeks. Treatments will be standardized; however, given the heterogeneity of symptoms, components of the treatments will be individualized to the participants based on what subgroup they're classified into at baseline based on their initial clinical examination and self-reported dominant impairment. Regardless of subgroup classification, as part of individualized care, all patients will receive reassurance and psychoeducation about the bio-psycho-social understanding of persistent symptoms, including advice on adaptive illness behaviours, such as gradually resuming premorbid activities and avoiding excessive rest and "all-or-nothing behaviour".
  Interventions: Other: Non-pharmacological Individualized rehabilitative therapy
- Usual care (Active Comparator): Active control - All participants in the active control group will receive 'usual care', (twice a week for 6 weeks), which will consist of reassurance and psychoeducation via the bio-psycho-social model on understanding persistent symptoms, including advice on adaptive illness behaviours, such as gradually resuming premorbid activities and avoiding excessive rest and "all-or-nothing behaviour". Additionally, participants will be afforded weekly 20-minute supervised progressive sub-symptom aerobic exercise sessions at the KITE clinic under the supervision of study coordinator. They will be instructed to also perform daily 20-minutes of subsymptom aerobic exercise outside the supervised exercise sessions.
  Interventions: Other: Non-pharmacological Usual care therapy

INTERVENTIONS:
Other: Non-pharmacological Individualized rehabilitative therapy — Treatments will be standardized but components of the treatments will be individualized to the participants based on what subgroup they're classified into at baseline based on their initial clinical examination and self-reported dominant impairment. *Physiological group - Participants will receive supervised sub-symptom aerobic exercise 20-minutes twice per week and mindfulness-based training 20-minutes twice per week. *Cervical group - Participants will receive physical therapy to the cervical spine. Physical therapy will include soft tissue therapy directed to the cervical myofascial tissues, and graded cervical spine facet mobilizations. *Vestibulo-Ocular group - Patients classified to vestibulo-ocular subgroup will receive bi-weekly 30-minute individualized oculomotor, vestibular and balance exercises including adaptation exercises, gaze stability exercises, visual-vestibular integration exercises, habituation exercises, static and dynamic balance exercises.
  Arms: Individualized care program
Other: Non-pharmacological Usual care therapy — All participants in the active control group will receive 'usual care', (twice a week for 6 weeks), which will consist of reassurance and psychoeducation via the bio-psycho-social model on understanding persistent symptoms, including advice on adaptive illness behaviours, such as gradually resuming premorbid activities and avoiding excessive rest and "all-or-nothing behaviour". Additionally, participants will be afforded weekly 20-minute supervised progressive sub-symptom aerobic exercise sessions at the KITE clinic under the supervision of study coordinator NM. They will be instructed to also perform daily 20-minutes of subsymptom aerobic exercise outside the supervised exercise sessions.
  Arms: Usual care

SUMMARY:
Protocol Summary

The present study was developed to better understand the effects and benefits of individualizing rehabilitative treatments based on subgroup classifications determined by a standardized clinical examination. The primary aim is to evaluate the response to individualized therapy on recovery, as measured by The Rivermead Post-concussion Symptoms Questionnaire (RPQ) and standardized clinical examination, when compared to an active control. The secondary aim is to evaluate the Pre and Post treatment state of the participants via a rapid advanced electroencephalography (EEG) when compared to the active control who will be provided the current standard form of therapy for persistent symptoms. The EEG changes will be compared to the standardized clinical examination findings as well as the RPQ.

Sample Size:

N= 50

Study Population

Participants will be eligible for study participation if they meet the following inclusion criteria: 21-years and older; diagnosed with postconcussion syndrome; and have adequate language skills in English to read and take part in rehabilitation treatment program. Participants will be excluded should: they have an unremarkable or normal clinical examination; have a chronic infectious disease; uncontrolled hypertension; other neurological disorders (not attributed to their primary diagnosis); cancer treatment (other than basal cell carcinoma), craniotomy, or refractory subdural hematoma long-term use of psychoactive medications that would compromise their ability to comprehend and perform study activities; those with pacemakers or elevated cardiovascular risk; ongoing litigation surrounding their injury; have been diagnosed with a moderate or severe brain injury prior to enrolment; post-concussive symptoms persisting beyond 12-months.

Study Design

The investigators will be conducting a 12-week case-crossover randomized controlled trial. Participants will undergo 6-weeks of care in their respective streams. After 6-weeks, participants will undergo a re-examination. They will then crossover and undertake the alternative treatment for 6-weeks. At the end of 12-weeks, participants will undertake the endpoint examinations.

Start Date:

May 2023

End Date:

September 2025

Primary Objective:

The primary aim is to evaluate the response to individualized therapy on recovery, as measured by The Rivermead Post-concussion Symptoms Questionnaire (RPQ) and standardized clinical examination, when compared to an active control.

DETAILED DESCRIPTION:
Background and Rationale

Disabilities secondary to traumatic brain injury are a major source of burden. Numerous treatments have been utilized and studied in an attempt to treat persistent postconcussive symptoms. However, the majority of clinical trials examined the efficacy of a single treatment. Given mild traumatic brain injury (mTBI) is a heterogenous condition characterized by a variety of clinical presentations, one could assume a lack of recovery or response to therapy when done in isolation.

The present study was developed to better understand the effects of individualized rehabilitative care in concussion patients. Specifically, the investigators seek to better understand the effects and benefits of individualizing rehabilitative treatments based on subgroup classifications determined by a standardized clinical examination. The investigators' intention is to establish a treatment methodology based on subgroup classification to individualized rehabilitative treatment programs. The primary aim is to evaluate the response to individualized therapy on recovery, as measured by The Rivermead Post-concussion Symptoms Questionnaire (RPQ) and standardized clinical examination, when compared to an active control. The secondary aim is to evaluate the Pre and Post treatment state of the participants via a rapid advanced EEG when compared to the active control who will be provided the current standard form of therapy for persistent symptoms. The electrophysiological changes will be compared to the standardized clinical examination findings as well as the RPQ.

Hypothesis

The investigators hypothesize that participants suffering from persistent post-concussive symptoms, with dominant somatic features, undergoing an individualized rehabilitation program derived from subgroup classification will demonstrate clinically meaningful and statistically significant improved RPQ scores when compared to the active control who will be provided the current standard form of therapy for persistent symptoms. Additionally, the investigators expect significantly improved brain vital sign as measured by rapid EEG, which will serve as a biomarker to confirm the clinical changes.

The investigators will be conducting a 12-week case-crossover randomized controlled trial. Participants will be randomized at baseline to either the individualized care program or an active control. No washout period will be used between interventions. It was assumed that given both interventional groups have a focus on rehabilitative therapy that no wash-out period was needed. Participants will undergo 6-weeks of care in their respective streams. After 6-weeks, participants will undergo a re-examination. They will then crossover and undertake the alternative treatment for 6-weeks. At the end of 12-weeks, participants will undertake the endpoint examinations.

ELIGIBILITY:
Inclusion Criteria:

* 21-years and older
* meet the definition of postconcussion syndrome, which requires a participant to report any 3 symptoms or more (from an inclusive list of 40 most commonly reported persisting symptoms) lasting at least 1-month following the diagnosis of a concussion. Concussion was defined according to the 5th International Consensus Statement on Concussion in Sport.
* Have adequate language skills in English to read and take part in rehabilitation treatment program.

Exclusion Criteria:

* In-patients at Toronto Rehabilitation Institute or any other affiliated University Health Network clinics.
* Participants will be excluded should their clinical examination be unremarkable for objective physical impairments,
* Have a chronic infectious disease,
* Uncontrolled hypertension,
* Other neurological disorders (not attributed to their primary diagnosis),
* Cancer treatment (other than basal cell carcinoma), craniotomy, or refractory subdural hematoma long-term use of psychoactive medications that would compromise their ability to comprehend and perform study activities, those with pacemakers or elevated cardiovascular risk,
* Ongoing litigation surrounding their injury,
* Have been diagnosed with a moderate or severe brain injury prior to enrolment, post-concussive symptoms persisting beyond 12-months.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2025-04-22 (Actual); Study Completion 2025-04-22 (Actual)

PRIMARY OUTCOMES:
Rivermead Postconcussion Questionnaire | Baseline; 6-weeks; 12-weeks
  The Rivermead Post-Concussion Symptom Questionnaire (RPQ) is a self-report scale to measure the severity of post-concussive symptoms following a Traumatic Brain Injury (TBI).
  Each item is rated on a 5-point ordinal scale: 0 = not experienced at all, 1 = no more of a problem, 2 = a mild problem, 3 = a moderate problem, and 4 = a severe problem. The total score is a sum of all items and ranges from 0 to 64 from (best to worst).

SECONDARY OUTCOMES:
Brain Vital Sign | Baseline; 6-weeks; 12-weeks
  Quantitative Electroencephalography (EEG). Brain vital sign as measured by rapid advanced electroencephalography (EEG) via NeuroCatchTM. NeuroCatch® conducts a rapid 6-minute scan to measure and report on three specific event related potentials (ERPs). ERPs are neurophysiological measures that are sensitive to changes in cognitive processing, which allows NeuroCatch® to assess an individual's cognitive brain health across various states. Specifically, the three ERPs, auditory N100 (auditory sensation); auditory oddball P300 (basic attention); and auditory speech processing N400 (cognitive processing) will be evaluated. Standardized normative data exists for all three ERP responses.
Patient Health Questionnaire (PHQ-9) | Baseline; 6-weeks; 12-weeks
  The Patient Health Questionnaire (PHQ) is an instrument used for making criteria-based diagnoses of depressive and other mental disorders commonly encountered in primary care. To score the instrument, the numbers of all the checked responses under each heading are tallied (not at all=0, several days=1, more than half the days=2, and nearly every day=3). There are nine items / questions scored from 0 = not at all, 1 = several days, 2 = more than half the days, 3 = nearly every day. The total score is a sum of all items and ranges from 0 to 27 (best to worst).
Neck Disability Index (NDI) | Baseline; 6-weeks; 12-weeks
  The Neck Disability Index (NDI) is a questionnaire designed to help us better understand how your neck pain affects your ability to manage everyday / life activities. The NDI has become a standard instrument for measuring self-rated disability due to neck pain and is used by both clinicians and researchers. Each of the 10 items scores from 0 to 5: 0 = no disability and 5 = complete. The maximum score is 50.

CONTACTS AND LOCATIONS:
Overall Officials: Milos R Popovic, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Rehabilitation Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with any other researchers.

REFERENCES:
- [Derived] Moser N, Popovic MR, Kalsi-Ryan S. Effectiveness of personalized rehabilitation in adults suffering from persistent concussion symptoms as compared to usual care: a randomized control trial protocol. BMC Neurol. 2024 Jul 10;24(1):239. doi: 10.1186/s12883-024-03700-5. PMID 38987676